CLINICAL TRIAL: NCT00971243
Title: A Phase IIb, Double-blind, Parallel Group, Multi-center, Dose-finding Study to Investigate the Efficacy and Safety of 4 Doses of MP-513 When Added to Ongoing Metformin Monotherapy in Subjects With Type 2 Diabetes Mellitus, With an Open Label Extension
Brief Title: Efficacy and Safety of MP-513 in Combination With Metformin in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MP-513-E07
Record Dates: First submitted 2009-09-01; First posted 2009-09-03 (Estimated); Results first posted 2014-09-01 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Insulin resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- MP-513 Lowest Dose and Metformin (Experimental)
  Interventions: Drug: MP-513 Lowest Dose and Metformin
- MP-513 Low Dose and Metformin (Experimental)
  Interventions: Drug: MP-513 Low Dose and Metformin
- MP-513 Medium Dose and Metformin (Experimental)
  Interventions: Drug: MP-513 Medium Dose and Metformin
- MP-513 High Dose and Metformin (Experimental)
  Interventions: Drug: MP-513 High Dose and Metformin
- Placebo and Metformin (Placebo Comparator)
  Interventions: Drug: Placebo and Metformin

INTERVENTIONS:
Drug: MP-513 Lowest Dose and Metformin — MP-513 tablets, once a day and Metformin tablets, for 24 weeks and extension treatment for up to 52 weeks.
  Arms: MP-513 Lowest Dose and Metformin
Drug: MP-513 Low Dose and Metformin — MP-513 tablets, once a day and Metformin tablets, for 24 weeks and extension treatment for up to 52 weeks.
  Arms: MP-513 Low Dose and Metformin
Drug: MP-513 Medium Dose and Metformin — MP-513 tablets, once a day and Metformin tablets, for 24 weeks and extension treatment for up to 52 weeks.
  Arms: MP-513 Medium Dose and Metformin
Drug: MP-513 High Dose and Metformin — MP-513 tablets, once a day and Metformin tablets, for 24 weeks and extension treatment for up to 52 weeks.
  Arms: MP-513 High Dose and Metformin
Drug: Placebo and Metformin — Placebo tablets once a day, and Metformin tablets, for 24 weeks and extension treatment for up to 52 weeks.
  Arms: Placebo and Metformin

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of MP-513 in combination with Metformin in patients with type 2 diabetes for 24 weeks administration and to evaluate the safety and efficacy of MP-513 in combination with Metformin with an extension treatment for up to 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are aged ≧ 18 years old.
* Patients whose HbA1c is ≧ 7.0 % and < 10.0%.
* Patients whose BMI is ≧ 20.0 and ≦40.0 ㎏/㎡.
* Patients who took metformin monotherapy for at least 56 consecutive days at the screening visit.

Exclusion Criteria:

* Patients with type 1 diabetes or secondary form of diabetes.
* Patients with heart failure symptoms.
* Patients with serious diabetic complications.
* Patients with severe hepatic disorder or severe renal disorder.
* Patients who are the excessive alcohol addicts.
* Patients who are pregnant, lactating and probably pregnant patients and patients who can not agree to contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 448 (Actual)
Dates: Start 2009-08; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Kerr, Dr, Principal Investigator — Royal Bournemouth Hospital
Locations (44):
- Denmark (3):
  - Aalborg
  - Ballerup Municipality
  - Vejle
- Germany (7):
  - Falkensee
  - Hamburg
  - Karlsruhe
  - Kiel
  - Ludwigshafen
  - Lübeck
  - Mainz
- Hungary (10):
  - Ádám
  - Békéscsaba
  - Budapest
  - Gyöngyös
  - Kaposvár
  - Miskolc
  - Nyíregyháza
  - Semmelweis
  - Szentes
  - Szigetvár
- Lithuania (3):
  - Kaunas
  - Klaipėda
  - Vilnius
- Poland (8):
  - Gdansk
  - Krakow
  - Leszno
  - Lodz
  - Niemodlin
  - Płock
  - Warsaw
  - Wroclaw
- Romania (6):
  - Brasov
  - Bucharest
  - Galati
  - Ploieşti
  - Timișoara
  - Timuș
- United Kingdom (7):
  - Addlestone
  - Ayr
  - Bournemouth
  - East Sussex
  - Edinburgh
  - Oldham
  - York

REFERENCES:
- [Derived] Kadowaki T, Kondo K. Efficacy and safety of teneligliptin added to glimepiride in Japanese patients with type 2 diabetes mellitus: a randomized, double-blind, placebo-controlled study with an open-label, long-term extension. Diabetes Obes Metab. 2014 May;16(5):418-25. doi: 10.1111/dom.12235. Epub 2013 Dec 10. PMID 24205974

RESULTS

PARTICIPANT FLOW:
Groups:
- Teneli 5mg+Met: Teneligliptin 5mg for 24 weeks (double-blind period) followed by teneligliptin20 mg for additional 28 weeks (open-label period) in combination with Metformin
- Teneli 10mg+Met: Teneligliptin 10mg for 24 weeks (double-blind period) followed by teneligliptin20 mg for additional 28 weeks (open-label period) in combination with Metformin
- Teneli 20mg+Met: Teneligliptin 20mg for 24 weeks (double-blind period) followed by teneligliptin20 mg for additional 28 weeks (open-label period) in combination with Metformin
- Teneli 40mg+Met: Teneligliptin 40mg for 24 weeks (double-blind period) followed by teneligliptin20 mg for additional 28 weeks (open-label period) in combination with Metformin
- Placebo+Met: Placebo for 24 weeks (double-blind period) followed by teneligliptin20 mg for additional 28 weeks (open-label period) in combination with Metformin
Period: Double Blind Period
Arm/Group | Teneli 5mg+Met | Teneli 10mg+Met | Teneli 20mg+Met | Teneli 40mg+Met | Placebo+Met
Started | 87 | 93 | 91 | 88 (One subject who did not receive any study drug was excluded from the ITT) | 88
Completed | 68 | 82 | 72 | 74 | 70
Not Completed | 19 | 11 | 19 | 14 | 18
Not completed — Adverse Event | 2 | 3 | 2 | 2 | 3
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0 | 1
Not completed — Physician Decision | 10 | 6 | 7 | 6 | 7
Not completed — Protocol Violation | 2 | 0 | 3 | 2 | 2
Not completed — Withdrawal by Subject | 4 | 1 | 4 | 4 | 4
Not completed — Other reasons | 1 | 0 | 2 | 0 | 1
Period: Open-label Period
Arm/Group | Teneli 5mg+Met | Teneli 10mg+Met | Teneli 20mg+Met | Teneli 40mg+Met | Placebo+Met
Started | 68 | 81 (One Subject did not entered because of the failure of inclusion/exclusion criteria.) | 71 (One Subject did not entered the Open-label Period because of the withdrawal of consent.) | 74 | 70
Completed | 60 | 71 | 66 | 64 | 64
Not Completed | 8 | 10 | 5 | 10 | 6
Not completed — Adverse Event | 1 | 0 | 1 | 1 | 0
Not completed — Physician Decision | 5 | 9 | 3 | 7 | 2
Not completed — Protocol Violation | 1 | 1 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 2 | 1
Not completed — Other reason | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Teneli 5mg+Met | Teneli 10mg+Met | Teneli 20mg+Met | Teneli 40mg+Met | Placebo+Met | Total
Number analyzed (Participants) | 87 | 93 | 91 | 88 | 88 | 447
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (7.7) | 58.5 (8.4) | 58.3 (9.5) | 58.2 (8.6) | 58.9 (8.2) | 58.5 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 42 | 35 | 36 | 41 | 195
  Male | 46 | 51 | 56 | 52 | 47 | 252

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline to Week 24
Description: The change of HbA1c from baseline to Week 24 or a last observation carried forward (LOCF), was assessed with an analysis of covariance (ANCOVA) model, with the centre and treatment effect as factors and the baseline HbA1c as a covariate.
Time Frame: Baseline and Week 24
Population: LOCF was implemented in the Intention-to-Treat (ITT) population analysis to replace missing values for all those subjects who did not present an HbA1c value at Week 24.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Teneli 5mg+Met | Teneli 10mg+Met | Teneli 20mg+Met | Teneli 40mg+Met | Placebo+Met
Number analyzed (Participants) | 87 | 93 | 91 | 88 | 88
percentage of HbA1c | -0.58 (0.07) | -0.68 (0.07) | -0.76 (0.07) | -0.91 (0.07) | -0.28 (0.07)

2. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) From Baseline to Week 24
Description: Change in FPG from baseline to Week 24 or LOCF was assessed with an ANCOVA approach similar to that of the primary efficacy endpoint.
Time Frame: Baseline and Week 24
Population: LOCF was implemented in the ITT population analysis to replace missing values for all those subjects who did not present a FPG value at Week 24.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Teneli 5mg+Met | Teneli 10mg+Met | Teneli 20mg+Met | Teneli 40mg+Met | Placebo+Met
Number analyzed (Participants) | 87 | 93 | 91 | 88 | 88
mg/dL | -15.54 (2.94) | -13.65 (2.83) | -17.84 (2.86) | -21.85 (2.91) | -3.51 (2.95)

3. Secondary Outcome: Adverse Events, Laboratory Tests, Vital Signs, Etc.
Time Frame: Weeks 24, 52
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 24 weeks
Groups:
- Teneli 5mg+Met: Teneligliptin 5mg plus Metformin
- Teneli 10 mg+Met: Teneligliptin 10mg plus Metformin
- Teneli 20 mg+Met: Teneligliptin 20mg plus Metformin
- Teneli 40 mg+Met: Teneligliptin 40mg plus Metformin
- Placebo+Met: Placebo plus Metformin
Arm/Group | Teneli 5mg+Met | Teneli 10 mg+Met | Teneli 20 mg+Met | Teneli 40 mg+Met | Placebo+Met
Serious Adverse Events (participants affected / at risk) | 4/87 | 4/93 | 3/91 | 5/88 | 6/88
Other Adverse Events (participants affected / at risk) | 43/87 | 43/93 | 41/91 | 36/88 | 48/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Teneli 5mg+Met (N=87) | Teneli 10 mg+Met (N=93) | Teneli 20 mg+Met (N=91) | Teneli 40 mg+Met (N=88) | Placebo+Met (N=88)
BRONCHITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1
PNEUMONIA (Infections and infestations) | 1 | 0 | 0 | 0 | 0
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
METASTASES TO LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
CEREBELLAR INFARCTION (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
IIIRD NERVE PARALYSIS (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
ISCHAEMIC STROKE (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
FEMORAL ARTERY OCCLUSION (Vascular disorders) | 0 | 1 | 0 | 0 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
MALLORY-WEISS SYNDROME (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
UMBILICAL HERNIA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
FATTY LIVER ALCOHOLIC (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
HEPATIC STEATOSIS (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Teneli 5mg+Met (N=87) | Teneli 10 mg+Met (N=93) | Teneli 20 mg+Met (N=91) | Teneli 40 mg+Met (N=88) | Placebo+Met (N=88)
BRONCHITIS (Infections and infestations) | 3 | 3 | 0 | 0 | 1
CYSTITIS (Infections and infestations) | 2 | 4 | 1 | 5 | 1
EAR INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 1
ERYSIPELAS (Infections and infestations) | 0 | 0 | 0 | 0 | 1
GASTROENTERITIS (Infections and infestations) | 1 | 0 | 1 | 3 | 2
GASTROENTERITIS VIRAL (Infections and infestations) | 1 | 0 | 0 | 0 | 0
HERPES SIMPLEX (Infections and infestations) | 1 | 0 | 0 | 0 | 0
INFLUENZA (Infections and infestations) | 1 | 1 | 0 | 0 | 0
LARYNGITIS (Infections and infestations) | 0 | 1 | 0 | 0 | 0
MEASLES (Infections and infestations) | 0 | 1 | 0 | 0 | 0
NASOPHARYNGITIS (Infections and infestations) | 6 | 4 | 2 | 7 | 6
ONYCHOMYCOSIS (Infections and infestations) | 0 | 0 | 1 | 0 | 0
OTITIS EXTERNA (Infections and infestations) | 0 | 0 | 1 | 0 | 0
PELVIC INFLAMMATORY DISEASE (Infections and infestations) | 0 | 0 | 0 | 1 | 0
PHARYNGITIS (Infections and infestations) | 1 | 0 | 0 | 1 | 2
PNEUMONIA (Infections and infestations) | 1 | 0 | 1 | 0 | 0
RASH PUSTULAR (Infections and infestations) | 1 | 0 | 0 | 0 | 0
SINUSITIS (Infections and infestations) | 1 | 0 | 1 | 0 | 1
TINEA PEDIS (Infections and infestations) | 0 | 1 | 0 | 0 | 0
TOOTH ABSCESS (Infections and infestations) | 0 | 1 | 0 | 0 | 0
TRACHEOBRONCHITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 1 | 3 | 0 | 2
URINARY TRACT INFECTION (Infections and infestations) | 2 | 3 | 2 | 0 | 2
VIRAL INFECTION (Infections and infestations) | 1 | 1 | 1 | 0 | 0
VULVAL ABSCESS (Infections and infestations) | 1 | 0 | 0 | 1 | 0
TOOTH INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | 0
ANAL ABSCESS (Infections and infestations) | 0 | 0 | 0 | 1 | 0
GINGIVAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 1
GENITOURINARY TRACT INFECTION (Infections and infestations) | 0 | 1 | 0 | 0 | 0
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 1 | 0 | 0 | 0 | 1
RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 0 | 0 | 1 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
MELANOCYTIC NAEVUS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
ANAEMIA (Blood and lymphatic system disorders) | 1 | 1 | 1 | 0 | 2
HYPOCHROMIC ANAEMIA (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
MICROCYTIC ANAEMIA (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
LYMPHATIC DISORDER (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
HYPOTHYROIDISM (Endocrine disorders) | 0 | 0 | 1 | 1 | 0
AUTOIMMUNE THYROIDITIS (Endocrine disorders) | 0 | 0 | 1 | 0 | 0
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
GOUT (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0 | 1
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 3 | 1 | 1
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 1 | 1 | 2 | 1
OBESITY (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
VITAMIN B12 DEFICIENCY (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
DYSLIPIDAEMIA (Metabolism and nutrition disorders) | 0 | 3 | 1 | 0 | 1
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
ANXIETY (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
CEREBRAL ATROPHY (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
DIABETIC NEUROPATHY (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
DIZZINESS (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
HEADACHE (Nervous system disorders) | 1 | 2 | 5 | 1 | 1
MEMORY IMPAIRMENT (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
MIGRAINE (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
SCIATICA (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
SYNCOPE (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
LACUNAR INFARCTION (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
CEREBROVASCULAR INSUFFICIENCY (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
CATARACT (Eye disorders) | 1 | 0 | 0 | 0 | 0
CONJUNCTIVITIS (Eye disorders) | 1 | 0 | 0 | 0 | 0
CONJUNCTIVITIS ALLERGIC (Eye disorders) | 0 | 0 | 0 | 0 | 1
DIABETIC RETINOPATHY (Eye disorders) | 1 | 1 | 0 | 0 | 0
EYE INFLAMMATION (Eye disorders) | 1 | 0 | 0 | 1 | 0
GLAUCOMA (Eye disorders) | 0 | 1 | 0 | 0 | 0
MACULAR DEGENERATION (Eye disorders) | 1 | 0 | 0 | 0 | 0
PERIORBITAL OEDEMA (Eye disorders) | 0 | 1 | 0 | 0 | 0
VERTIGO (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 2
ANGINA PECTORIS (Cardiac disorders) | 0 | 1 | 2 | 0 | 0
AORTIC VALVE SCLEROSIS (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 1 | 0 | 1 | 1
ATRIOVENTRICULAR BLOCK FIRST DEGREE (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
CARDIAC FAILURE (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
CARDIOMYOPATHY (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
HYPERTENSIVE HEART DISEASE (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
LEFT VENTRICULAR FAILURE (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
SINUS BRADYCARDIA (Cardiac disorders) | 0 | 2 | 0 | 0 | 0
TACHYCARDIA (Cardiac disorders) | 0 | 2 | 0 | 0 | 0
MITRAL VALVE SCLEROSIS (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
FLUSHING (Vascular disorders) | 1 | 0 | 0 | 0 | 0
HYPERTENSION (Vascular disorders) | 5 | 2 | 3 | 2 | 2
VARICOSE ULCERATION (Vascular disorders) | 0 | 0 | 1 | 0 | 0
VENOUS INSUFFICIENCY (Vascular disorders) | 0 | 1 | 0 | 0 | 0
HOT FLUSH (Vascular disorders) | 0 | 0 | 1 | 1 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 1 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
VASOMOTOR RHINITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 1 | 2 | 5 | 1 | 3
DRY MOUTH (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
DYSPEPSIA (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0
FLATULENCE (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
GASTRITIS EROSIVE (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
GINGIVITIS (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 1
REFLUX OESOPHAGITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
VOMITING (Gastrointestinal disorders) | 1 | 2 | 1 | 1 | 0
ABDOMINAL HERNIA (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
APICAL GRANULOMA (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
HEPATIC STEATOSIS (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 2
ACTINIC KERATOSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
CUTANEOUS SARCOIDOSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
DERMAL CYST (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
ECZEMA (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 2
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0
HYPERKERATOSIS (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
INGROWING NAIL (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 2
RASH (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0 | 0
RASH VESICULAR (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
SKIN FISSURES (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
ONYCHOCLASIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
PHOTODERMATOSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 2
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 1
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
HAEMARTHROSIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
JOINT EFFUSION (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 2
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
SYNOVITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
TENOSYNOVITIS STENOSANS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
FOOT DEFORMITY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
GLYCOSURIA (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1
MICROALBUMINURIA (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
POLLAKIURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
RENAL COLIC (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
RENAL FAILURE CHRONIC (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
DIABETIC NEPHROPATHY (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1
STRESS URINARY INCONTINENCE (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
EPIDIDYMITIS (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | 0
OVARIAN CYST (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
CHEST PAIN (General disorders) | 0 | 1 | 1 | 1 | 2
FATIGUE (General disorders) | 0 | 0 | 0 | 2 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 0 | 0 | 1 | 0 | 0
MALAISE (General disorders) | 0 | 0 | 0 | 0 | 1
OEDEMA PERIPHERAL (General disorders) | 1 | 0 | 0 | 1 | 0
PAIN (General disorders) | 0 | 1 | 0 | 0 | 0
PYREXIA (General disorders) | 0 | 1 | 0 | 0 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0 | 0 | 2 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 1 | 0 | 0
BLOOD CHOLESTEROL INCREASED (Investigations) | 0 | 1 | 0 | 0 | 0
BLOOD CREATININE INCREASED (Investigations) | 0 | 0 | 1 | 0 | 0
BLOOD PRESSURE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 1
BLOOD TRIGLYCERIDES INCREASED (Investigations) | 2 | 1 | 0 | 1 | 0
BLOOD UREA INCREASED (Investigations) | 1 | 0 | 0 | 0 | 0
C-REACTIVE PROTEIN INCREASED (Investigations) | 1 | 2 | 2 | 1 | 0
CREATININE RENAL CLEARANCE DECREASED (Investigations) | 0 | 0 | 1 | 0 | 0
CRYSTAL URINE PRESENT (Investigations) | 0 | 0 | 1 | 0 | 0
HEART RATE IRREGULAR (Investigations) | 0 | 0 | 0 | 0 | 1
LIVER FUNCTION TEST ABNORMAL (Investigations) | 1 | 0 | 0 | 0 | 0
WEIGHT DECREASED (Investigations) | 1 | 0 | 0 | 0 | 0
PROTEIN URINE PRESENT (Investigations) | 0 | 0 | 1 | 1 | 0
URINE URIC ACID INCREASED (Investigations) | 1 | 0 | 0 | 0 | 0
HEPATIC ENZYME INCREASED (Investigations) | 0 | 2 | 0 | 0 | 1
HAND FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
SOFT TISSUE INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
TENDON RUPTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
CONTUSION (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
SKIN LACERATION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
OPEN WOUND (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0
LIGAMENT INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
LIMB INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
ORCHIDECTOMY (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other